CLINICAL TRIAL: NCT07076888
Title: Impact of Aerobic Exercises on Serum Uric Acid Levels in Hemodialysis Patients
Brief Title: Aerobic Exercises and Hemodialysis Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Doaa Rafat, Assistant Professor of Physical Therapy, Faculty of Physical Therapy, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/025/00123
Record Dates: First submitted 2025-06-10; First posted 2025-07-22 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Hemodialysis
Keywords: Aerobic exercise; hemodialysis; serum uric acid; quality of life
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Group A (study Group): 16 HD patients received a conventional physical therapy program (breathing, stretching, and lower limb circulatory exercises) combined with the aerobic exercise program.
  Interventions: Other: Aerobic Exercises; Other: Conventional Program
- Group B (Active Comparator): Group B (Control Group): 16 HD patients received only the conventional physical therapy program.
  Interventions: Other: Conventional Program

INTERVENTIONS:
Other: Aerobic Exercises — 1. Timing of Exercise:
     Aerobic exercises were performed on non-dialysis days. This scheduling avoids post-dialysis fatigue and hypotensive effects, optimizing patient safety and performance.
  2. Frequency:
     Patients was engaged in aerobic exercise 3 times per week on non-consecutive days, to allow sufficient recovery time between sessions.
  3. Duration of Each Session:
     * Total Duration: Each exercise session was last between 20 to 45 minutes.
     * Warm-Up: 5-10 minutes of low-intensity activity (e.g., slow walking).
     * Main Exercise: 15-30 minutes of moderate-intensity aerobic exercise.
     * Cool-Down:*5-10 minutes of gradual reduction in intensity.
  4. Exercise Modality:
     * Options: Patients may choose between treadmill walking or using a stationary bike, depending on their preference, physical condition.
     * Variety: To maintain engagement and reduce monotony, patients can alternate between treadmill and bike exercises.
  5. Intensity:
  Use moderate-intensity exercise, aiming for 60-70% of the p
  Arms: Group A
Other: Conventional Program — 1. Breathing Exercises
  - Diaphragmatic Breathing: Instruct patients to place one hand on their chest and the other on their abdomen. They should inhale deeply through their nose, allowing the abdomen to rise, and then exhale slowly through their mouth. This breathing technique has been shown to reduce stress, improve respiratory efficiency, and enhance relaxation . For optimal benefits, patients should practice this for 5-10 minutes, 2-3 times a day.
  Stretching Exercises Hamstring Stretch: Instruct patients to sit with one leg extended straight out in front of them and the other leg bent. They should reach towards the toes of the extended leg while keeping their back straight. Hold the stretch for 20-30 seconds and repeat the stretch 2-3 times per leg.
  Lower Limb Circulatory Exercises Ankle Pumps: While lying down or seated, instruct patients to alternately point and flex their feet to stimulate circulation and improve lower leg mobility. Perform 20-30 pumps per foot, 2-3 times a day

SUMMARY:
Patients undergoing hemodialysis (HD) frequently exhibit elevated serum uric acid (SUA) levels, which are associated with cardiovascular risks, joint issues, and diminished quality of life (QoL). Aerobic exercise has been shown to improve cardiovascular health and reduce SUA levels in various populations, suggesting potential benefits for HD patients.

Objective: This study aimed to investigate the impact of aerobic exercise on serum uric acid (SUA) levels, functional capacity, and quality of life (QoL) in patients undergoing hemodialysis (HD).

Methods: This randomized controlled trial will recruit 32 participants, aged 40-60, undergoing HD. The intervention group (Group A) will participate in a structured 6-week aerobic exercise program, while the control group (Group B) will receive only conventional physical therapy. Pre- and post-intervention assessments included SUA levels, the Six-Minute Walk Test (6MWT), and the Kidney Disease Quality of Life Short Form (KDQOL-SF™)

DETAILED DESCRIPTION:
32 Subjects of both genders will participate in this study at El-khazendara Hospitals with age ranged between (40-60) years old. They will receive a comprehensive verbal and written explanation of the study, including its objectives, procedures, and potential benefits.

participants will randomly assigned into two equal groups using a sealed-envelope randomization method to ensure unbiased allocation.

* Group A (study Group): 16 HD patients receiving a conventional physical therapy program (breathing, stretching, and lower limb circulatory exercises) plus the aerobic exercise program.
* Group B (Control Group): 16 HD patients receiving only the conventional physical therapy program.

  6-weeks of aerobic exercise program (3 sessions per week, 20-45 minutes each session)

Outcome measures include:

* Serum Uric Acid: Measured using an automated biochemistry analyzer, with results reported in mg/dL.
* Functional Capacity: Assessed using the Six-Minute Walk Test (6MWT), a validated tool used to evaluate exercise tolerance and endurance in clinical populations.
* Quality of Life:Measured using the Kidney Disease Quality of Life Short Form (KDQOL-SF™) Arabic Version, which assesses various domains related to both physical and mental health.

ELIGIBILITY:
Inclusion Criteria:

1. Hemodialysis patients aged 40-60years
2. Patients are medically stable and able to participate in physical activity.
3. Participants are able to understand the commands.
4. Participants must be stable on hemodialysis for at least 3 months.

Exclusion Criteria:

1. Patients with significant cardiovascular or respiratory diseases, or other conditions that could impair their ability to exercise.
2. Severe cognitive impairment or psychiatric conditions that could interfere with study participation.
3. patients with acute medical conditions.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Serum Uric Acid | from enrollment to the end of 6 weeks of treatment

SECONDARY OUTCOMES:
Change in Functional ability of the patient | from enrollment to the end of 6 weeks of treatment
  Assessed by using the Six-Minute Walk Test (6MWT), a validated tool used to evaluate exercise tolerance and endurance in clinical populations.
Change in Quality of life | from enrollment to the end of 6 weeks of treatment
  Kidney Disease Quality of Life Short Form (KDQOL-SF™): The KDQOL-SF™ is a key tool used to assess the quality of life in patients with chronic kidney disease, particularly those undergoing hemodialysis. This version of the questionnaire measures multiple domains, including physical functioning, emotional well-being, and social roles, with a focus on issues specific to kidney disease such as symptoms, work status, and patient satisfaction. The scores are transformed into a scale from 0 to 100, with higher scores indicating a better quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Heba Elfeky Lecturer of physical therapy - Cairo University, lecturer, Study Director — Department of Basic sciences for physical therapy, Faculty of Physical Therapy , Cairo university, Cairo, Egypt
Locations (1):
- Physical Therapy faculty, Cairo University, Cairo, Egypt